CLINICAL TRIAL: NCT00477113
Title: TYGRIS: TYSABRI® Global Observational Program in Safety
Brief Title: TYSABRI Global Observational Program in Safety
Acronym: TYGRIS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS402
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Sclerosis
Keywords: natalizumab; MS; Tysabri; Multiple Sclerosis; TYGRIS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The Primary objective of this study is to determine the incidence and pattern of serious infections, malignancies, and other serious adverse events (SAE) in participants with multiple sclerosis (MS) treated with Tysabri (natalizumab).

DETAILED DESCRIPTION:
The TYSABRI Global Observational Program in Safety (TYGRIS) is a safety observational cohort program designed to obtain long-term safety data in multiple sclerosis (MS) participants treated with natalizumab in a clinical practice setting in the United States or Canada.

ELIGIBILITY:
Key Inclusion Criteria:

* MS patients in the US and Canada receiving TYSABRI under standard clinical care for less than or equal to 3 infusions are eligible to participate in TYGRIS.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MS patients treated with TYSABRI in North America
Sampling Method: Non-Probability Sample
Enrollment: 2207 (Actual)
Dates: Start 2007-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious infections, malignancies, and other SAEs | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- There may be mulitple sites in this clinical trial. Contact United BioSource Corporation, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Foley J, Carrillo-Infante C, Smith J, Evans K, Ho PR, Lee L, Kasliwal R, Stangel M, Vermersch P, Hutchinson M, Marinelli F, Smirnakis K; TYGRIS investigators. The 5-year Tysabri global observational program in safety (TYGRIS) study confirms the long-term safety profile of natalizumab treatment in multiple sclerosis. Mult Scler Relat Disord. 2020 Apr;39:101863. doi: 10.1016/j.msard.2019.101863. Epub 2019 Nov 21. PMID 31901758
- See also: TYGRIS US Home Page — https://www.tygris.com/public/default.aspx